CLINICAL TRIAL: NCT01159925
Title: Epidemiologic Surveillance to Assess Trends in Acute Hepatitis A Among Children in Panama
Brief Title: Surveillance Study to Determine the Trends in Acute Hepatitis A Among Panamanian Children
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112158
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Acute Hepatitis A; Hepatitis
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum

GROUPS / COHORTS (3):
- Possible hepatitis A Cohort: Children with an acute disease characterized by discrete onset of symptoms and jaundice
  Interventions: Procedure: Serum sample
- Probable hepatitis A Cohort: Children with an increase in serum levels of transaminase 2.5 times higher than the maximum limit of the normal interval
  Interventions: Procedure: Serum sample
- Confirmed hepatitis A Cohort: Children presenting a positive result for Immunoglobulin M for hepatitis A virus
  Interventions: Procedure: Serum sample

INTERVENTIONS:
Procedure: Serum sample — Serum samples collected

SUMMARY:
The purpose of this study is to collect epidemiological and clinical data to assess the vaccine impact and occurrence of confirmed acute hepatitis A cases in sentinel hospitals after the introduction of Havrix™ into the Expanded Program of Immunization.

DETAILED DESCRIPTION:
This is an observational, prospective, multi-centre, sentinel based study in 3 hospitals in Panama. Hospitals are selected based on population density or hepatitis A disease burden.

The Pan American Health Organization (PAHO) definition for a possible case of acute hepatitis A are used for subjects aged between >1 month and <15 years.

Data regarding clinical and epidemiologic information are collected and serum samples are collected to test hepatitis A markers and determine if infection with hepatitis A virus has recently occurred.

Surveillance will be for a period of approximately 2.5 years from the date of study initiation.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between >1 month and <15 years of age at the time of enrolment, being referred to any of the 3 participating sentinel hospitals.
* Subjects with clinical diagnosis of possible acute hepatitis A.
* Written informed consent obtained from the parent or guardian of the subject.
* Subjects for whom a blood sample is collected.

Exclusion Criteria:

* Subjects with confirmed diagnosis of non-viral hepatitis

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged >1 month and <15 years of age being seen for possible acute hepatitis A during the study time period at the selected sentinel hospitals of Panama
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of confirmed acute hepatitis A cases identified in the selected sentinel hospitals during the study period by age group, area of residence and year of surveillance | average time-frame: 2.5 years

SECONDARY OUTCOMES:
Occurrence of possible and probable cases of acute hepatitis A virus by age group, area of residence and year of surveillance | average time-frame: 2.5 years
Risk factors for confirmed cases of acute hepatitis A | average time-frame: 2.5 years
Frequency of different clinical signs and symptoms of hepatitis A | average time-frame: 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Clayton, Provincia de Panamá, Panama

REFERENCES:
- [Derived] Estripeaut D, Contreras R, Tinajeros O, Castrejon MM, Shafi F, Ortega-Barria E, DeAntonio R. Impact of Hepatitis A vaccination with a two-dose schedule in Panama: Results of epidemiological surveillance and time trend analysis. Vaccine. 2015 Jun 22;33(28):3200-7. doi: 10.1016/j.vaccine.2015.04.100. Epub 2015 May 14. PMID 25981490